CLINICAL TRIAL: NCT03717038
Title: A Phase 3, Randomized, Open-Label, Multicenter Trial of Sym004 Versus Trifluridine/Tipiracil (TAS-102) in Patients With Chemotherapy-Refractory or Relapsed Metastatic Colorectal Carcinoma and Acquired Resistance to Anti-EGFR Monoclonal Antibody Therapy
Brief Title: Sym004 Versus TAS-102 in Patients With mCRC
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was withdrawn due to administrative reasons
Sponsor: Symphogen A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sym004-12; 2018-003187-31 (EudraCT Number)
Record Dates: First submitted 2018-10-18; First posted 2018-10-23 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Metastatic Colorectal Cancer; Colorectal Cancer Metastatic; Carcinoma
Keywords: Metastatic Colorectal Cancer; Colorectal Cancer Metastatic; Carcinoma; Sym004; futuximab; modotuximab; TAS-102; Trifluridine; Tipiracil; Lonsurf
MeSH Terms: conditions — Colorectal Neoplasms; Carcinoma | interventions — futuximab; trifluridine tipiracil drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Sym004) (Experimental): Sym004 will be administered as a loading dose of 9 mg/kg on Cycle 1 Day 1, followed by weekly doses of 6 mg/kg beginning Cycle 1 Day 8.
  Interventions: Drug: Sym004
- Arm B (TAS-102) (Active Comparator): TAS-102 is commercially available and will be administered as per local prescribing instructions.
  Interventions: Drug: TAS-102

INTERVENTIONS:
Drug: Sym004 — Sym004 is a 1:1 mixture of two recombinant mAbs (futuximab and modotuximab) which bind specifically to non-overlapping epitopes located in the extracellular domain (ECD) of the EGFR.
  Arms: Arm A (Sym004)
Drug: TAS-102 — TAS-102 is a combination of trifluridine, a thymidine-based nucleic acid analogue, and tipiracil, a thymidine phosphorylase inhibitor.
  Other Names: Trifluridine/Tipiracil; Lonsurf
  Arms: Arm B (TAS-102)

SUMMARY:
This is a Phase 3, randomized, open-label, 2-arm trial designed to evaluate overall survival (OS) following treatment with Sym004, an investigational medicinal product (IMP), versus TAS-102 (trifluridine/tipiracil), a comparator (control) agent.

DETAILED DESCRIPTION:
Randomization is in the ratio of 1:1 to either Sym004 (Arm A) or TAS-102 (Arm B) in genomically-selected patients with chemotherapy-refractory or relapsed metastatic colorectal carcinoma (mCRC) and acquired resistance to anti-epidermal growth factor receptor (EGFR) monoclonal antibody (mAb) therapy.

Following consent, centralized genomic analysis will be conducted on blood samples obtained from each potential patient. Double-negative (DN) results as defined in trial inclusion criteria will be required for initial eligibility prior to randomization. Patients with DNmCRC will continue in the screening process. Once deemed fully eligible, patients will be randomized to either Arm A or Arm B (collectively referred to as protocol therapy).

Dosing cycles of 28 days with the assigned protocol therapy will continue until a protocol-specified discontinuation criterion is met. Following treatment discontinuation, patients will continue to be followed for OS.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, ≥ 18 years of age (≥ 20 years of age in Japan) at the time of obtaining informed consent.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1 (or equivalent Karnofsky PS of 70% to 100%).
* Histologically or cytologically confirmed adenocarcinoma of the colon or rectum that is metastatic.
* Meeting the protocol definition of DNmCRC as assessed in the screening blood test.
* mCRC not amenable to surgical intervention due to either medical contraindications or non-resectability of the tumor.
* Measurable or non-measurable disease according to the Response Evaluation Criteria in Solid Tumors (Version 1.1) (RECIST v1.1).
* Must have received ≥ 2 prior regimens of standard therapy for mCRC, or 1 prior regimen of standard adjuvant therapy and ≥ 1 prior regimen of standard therapy for mCRC, with failure of those regimens (due to refractory, relapsed, or progressive disease [PD], or due to intolerance warranting discontinuation and precluding retreatment with the same agent prior to PD). If one of the regimens utilized for inclusion is adjuvant therapy, the patient must have experienced documented recurrence by imaging studies within ≤ 6 months of completion of that therapy. Prior standard chemotherapy must have included agents as specified in the protocol (where approved in the country).
* Persons of childbearing potential agreeing to use a highly effective method of contraception during the study, beginning within 2 weeks prior to the first dose of protocol therapy and continuing until 3 months after the last dose of Sym004 or 6 months after the last dose of TAS-102; male patients must also agree to refrain from sperm donation during these periods.

Exclusion Criteria:

* Women who are pregnant or intending to become pregnant before, during, or within 3 months after the last dose of Sym004 or 6 months after the last dose of TAS-102; women who are breastfeeding.
* Prior history of specific mutations (specified in the protocol) in the tumor tissue at the time of any previous assessment.
* Known, untreated central nervous system (CNS) or leptomeningeal metastases, or spinal cord compression; patients with any of these not controlled by prior surgery or radiotherapy, or patients with symptoms suggesting CNS involvement for which treatment is required.
* An active second malignancy or history of another malignancy within 5 years prior to randomization, with exceptions.
* Active thrombosis, or a history of deep vein thrombosis or pulmonary embolism, within 4 weeks prior to randomization, unless adequately treated and considered by the Investigator to be stable.
* Active uncontrolled bleeding or a known bleeding diathesis.
* Known clinically significant cardiovascular disease or condition.
* Non-healing wounds on any part of the body.
* Significant gastrointestinal abnormality.
* Skin rash of Grade > 1 from prior anti-EGFR or other therapy at the time of randomization.
* Any other unresolved Grade > 1 toxicity associated with prior antineoplastic therapy, with exceptions.
* Known or suspected hypersensitivity to any of the excipients of formulated Sym004 or TAS-102.

Drugs and Other Treatments Exclusion Criteria:

* Prior treatment with either TAS-102 or regorafenib.
* Antineoplastic agents for the primary malignancy (standard or investigational) within 3 weeks prior to randomization and during study; includes chemotherapy, immunotherapy, or other biological therapy.
* Other investigational treatments within 3 weeks prior to randomization and during study; includes participation in medical device or other therapeutic intervention clinical trial.
* Radiotherapy within 3 weeks prior to randomization.
* Immunosuppressive or glucocorticoid therapy (> 10 mg daily prednisone or equivalent), within 2 weeks prior to randomization and during study; includes systemic or enteric corticosteroids.
* Prophylactic use of hematopoietic growth factors within 1 week prior to randomization and during Cycle 1 of study; thereafter prophylactic use of growth factors is allowed as clinically indicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-02 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) time following treatment with Sym004 versus TAS-102. | Assessed up to 5 years.
  Time (in months) from the date of randomization to the date of death. In the absence of death confirmation or for patients alive as of the OS data cut-off date (i.e., date upon reaching 445 deaths), OS will be censored at the date of last study follow-up, or the cut-off date, whichever is earlier.

SECONDARY OUTCOMES:
Antineoplastic Efficacy: Progression Free Survival (PFS) as assessed by Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST v1.1) | Assessed up to 5 years.
  Time (in months) from the date of randomization until the date of the investigator-assessed radiological disease progression or death due to any cause.
  Investigator-assessed radiological disease progression (per RECIST v1.1) with the following key censoring rules:
  * Patients who are alive with no disease progression as of the analysis cut-off date will be censored at the date of the last tumor assessment.
  * Patients who receive non-study cancer treatment before disease progression will be censored at the date of the last evaluable tumor assessment before the initiation of non-study cancer treatment.
  * Patients with clinical, but not radiologic, evidence of progression will be censored at the date of the last evaluable tumor assessment before the clinical progression assessment.
Antineoplastic Efficacy: Objective Response Rate (ORR) as assessed by RECIST v1.1. | Assessed up to 5 years.
  Defined as the proportion of patients with objective evidence of complete response (CR) or partial response (PR). Assessed approximately every 8 weeks (at the end of even-numbered cycles).
Antineoplastic Efficacy: Disease Control Rate (DCR) as assessed by RECIST v1.1. | Assessed up to 5 years.
  Defined as the proportion of patients with objective evidence of CR, PR, or stable disease (SD). Assessed approximately every 8 weeks (at the end of even-numbered cycles).
Antineoplastic Efficacy: Duration of Response (DOR) as assessed by RECIST v1.1. | Assessed up to 5 years.
  Time (in months) from the first documentation of response (CR or PR) to the first documentation of objective tumor progression or to death due to any cause, with the same censoring rules as for PFS.
Sym004 Safety Evaluation: Occurrence and nature of adverse events (AEs) on a weekly dosing regimen. | Assessed up to 5 years.
  AEs will be coded according to the Medical Dictionary for Regulatory Activities (MedDRA) terminology and the severity of the toxicities will be graded according to the Common Terminology Criteria for Adverse Events (Version 5) (CTCAE v5), where applicable, from signing of informed consent up to 30 days after the final dose of Sym004.
Immunogenicity Assessment: Number of subjects with anti-drug antibodies (ADAs) to Sym004 over time. | Assessed up to 5 years.
  Serum sampling to assess the potential for ADA formation are planned on the following visits: Cycle 1 Day 1, Cycle 1 Day 15, Cycle 2 Day 1, Day 1 of odd numbered cycles thereafter, the End of Treatment Visit, and the 1-Month Follow-up Visit.
Pharmacokinetic (PK) Parameters of Sym004: Trough Concentration (Cmin) | Assessed up to 5 years.
  Cmin is defined as the serum concentration at the start of infusion. The serum concentration of Sym004 is the sum of the two constituting mAbs, futuximab and modotuximab. Sparse sampling at 7 timepoints are planned on the following visits: Cycle 1 Day 1, Cycle 1 Day 8, Cycle 2 Day 1, Cycle 3 Day 1, End of Treatment Visit.
Pharmacokinetic (PK) Parameters of Sym004: Maximum Concentration (Cmax) | Assessed up to 5 years.
  Cmax is defined as the serum concentration at the end of infusion. The serum concentration of Sym004 is the sum of the two constituting mAbs, futuximab and modotuximab. Sparse sampling at 7 timepoints are planned on the following visits: Cycle 1 Day 1, Cycle 1 Day 8, Cycle 2 Day 1, Cycle 3 Day 1, End of Treatment Visit.

CONTACTS AND LOCATIONS:
Overall Officials: Josep Tabernero, MD, PhD, Principal Investigator — Vall d'Hebron Institute of Oncology (VHIO)

IPD SHARING:
Plan to Share IPD: Undecided